CLINICAL TRIAL: NCT00413621
Title: MRI of Alzheimer's Disease Imaging Amyloid Plaques in Persons With and Without Memory Problems
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070050; 07-N-0050
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-07

CONDITIONS: Alzheimer's Disease
Keywords: MRI; Alzheimer Disease; Amyloid; AD; Healthy Volunteer; HV
MeSH Terms: conditions — Alzheimer Disease

SUMMARY:
The study will investigate the possibility of detecting early signs of Alzheimer's disease using magnetic resonance imaging (MRI). If plaques, types of damage, can be imaged by MRI, the procedure could be used in clinical trials and may also help in the clinical diagnosis of patients. Alzheimer's disease, a progressive disease, is a major cause of functional disability and institutionalization, affecting 4.5 million people in the United States, a number that will more than triple by 2030 as the population ages.

Patients ages 55 to 90 who have mild symptoms of Alzheimer's disease and who are in good health may be eligible for this study. Twenty patients will be recruited from Johns Hopkins' Alzheimer's Disease Research Center. There will also be a control group of 20 people without the disease.

Healthy patients and volunteers will have a clinical MRI brain scan and a neurological examination at Johns Hopkins Hospital before the 7T MRI scan. Also, patients will have a Mini-Mental State Examination, a standardized test to evaluate memory, done at Johns Hopkins within 4 weeks of the 7T MRI. This study uses a device situated at the NIH Bethesda campus that operates at a high magnetic field strength of 7 Tesla, that is, the unit used to measure the strength of a strong magnet. The Food and Drug Administration has categorized MRI up to 8 Tesla as not a significant health risk. MRI scanning is routinely done at magnetic field strengths up to 4T. MRI images are created through the use of a large magnet and radio waves. During the procedure, patients lie on a table moved into a strong magnetic field. They are asked to lie still but can easily hear and speak to research staff. A respiratory belt is placed around the chest, and a finger probe is placed on the finger, to monitor breathing and heart rate. For obtaining a better picture, a special lightweight coil may be placed on or around the patient's head. The scan takes from 20 minutes to 2 hours, with most scans at 45 to 90 minutes. Due to limited experience with the use of 7T MRI and its investigational nature, patients will be asked to complete a questionnaire immediately after the study. They will be asked about their comfort level and if they experienced unusual sensations. Answers will be reviewed with patients by an experienced MRI investigator to get details of any unusual sensations reported. If patients experience unusual sensations, they are followed up by phone within 24 hours.

This study wi...

DETAILED DESCRIPTION:
Objective:

The objective of the proposed pilot study is to investigate the possibility of detecting early signs of Alzheimer's Disease (AD) using high field (7T) MRI. If plaques can be imaged by MRI, the procedure could be used as a measure of efficacy in clinical trials of AD, and replace more invasive methods such as positron emission tomography (PET). This procedure might also be helpful in the clinical diagnosis of patients.

Study Population:

The target population is a group of 20 Alzheimer's patients with mild cognitive impairment. As reference, an age-matched control group (n=20) will be recruited from the normal adult population.

Design:

Our working hypothesis is that high resolution MRI at 7T allows detection of amyloid plaques in AD. To test this hypothesis, subjects from AD and control population will each undergo an MRI at 7T to image brain structure at high resolution. Brain cortical structures will then be compared between the two groups and investigated for abnormalities.

Outcome Measure:

As outcome measure of this study, it will be determined if (sub) cortical plaques typical of AD are detectable with high field MRI.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any neurologically and psychiatrically normal, male or female, healthy volunteer ages 55-90 years old. Participants must be capable of understanding the procedures and requirements of this study and subjects must be willing to sign an informed consent document. Normal controls will demonstrate normal function in daily life, based on the Clinical Dementia Rating Scale (CDR). The CDR is administered annually to all JHADRC participants.
* AD patients will be required to meet the NINCDS/ADRDA criteria for AD. All patients must be mildly impaired. Severity will be measured by the Mini-Mental State Exam (MMSE) and only patients with an MMSE score of 20 - 26 will be included. They must be able to give informed consent.

EXCLUSION CRITERIA:

* Inability to cooperate.
* A subject will be excluded if he/she has a contraindication to MR scanning such as the following: claustrophobia, pregnancy, aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body (e.g. metal shavings) or insulin pump.
* Subjects who underwent brain surgery, or other neurological disease (e.g., stroke, Parkinson's disease, significant brain vascular disease, brain trauma).
* Evidence of cerebrovascular risk factors, including diabetes, arrhythmias, and lacunar infarcts seen on MRI.
* History of vertigo, seizure disorder, middle-ear disorder, and double vision.
* Active major psychiatric illness.
* Dental work such as ferromagnetic crowns or bridges.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-12-14; Primary Completion 2009-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Ferri CP, Prince M, Brayne C, Brodaty H, Fratiglioni L, Ganguli M, Hall K, Hasegawa K, Hendrie H, Huang Y, Jorm A, Mathers C, Menezes PR, Rimmer E, Scazufca M; Alzheimer's Disease International. Global prevalence of dementia: a Delphi consensus study. Lancet. 2005 Dec 17;366(9503):2112-7. doi: 10.1016/S0140-6736(05)67889-0. PMID 16360788
- [Background] Hebert LE, Scherr PA, Bienias JL, Bennett DA, Evans DA. Alzheimer disease in the US population: prevalence estimates using the 2000 census. Arch Neurol. 2003 Aug;60(8):1119-22. doi: 10.1001/archneur.60.8.1119. PMID 12925369
- [Background] Breitner JC, Wyse BW, Anthony JC, Welsh-Bohmer KA, Steffens DC, Norton MC, Tschanz JT, Plassman BL, Meyer MR, Skoog I, Khachaturian A. APOE-epsilon4 count predicts age when prevalence of AD increases, then declines: the Cache County Study. Neurology. 1999 Jul 22;53(2):321-31. doi: 10.1212/wnl.53.2.321. PMID 10430421